CLINICAL TRIAL: NCT05466253
Title: Effects of Early Versus Delayed Orthodontic Treatment After Periodontal Surgery on Periodontal Health in Periodontally Compromised Patients - a Randomized Clinical Trial
Brief Title: Early Versus Delayed Orthodontic Treatment After Periodontal Surgery on Periodontal Health in Periodontally Compromised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/21/20/ANUNAY
Record Dates: First submitted 2022-06-20; First posted 2022-07-20 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis, Adult
Keywords: ORTHODONTIC PERIODONTAL MANAGEMENT
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: All the patients included in the study will receive a detailed periodontal evaluation and all periodontal parameters (osseous and non-osseous) will be recorded at the baseline and Phase I periodontal therapy will be provided. This will include oral hygiene instruction, scaling and root planning and re-evaluation after one weeks. If the patients are able to maintain oral hygiene after preliminary periodontal intervention they will be included in further stages of the study. All the patients will receive the indicated periodontal surgical treatment. and the patients will then be randomly divided into two groups - test group and control group Orthodontic treatment will be started in the test group 10 days after periodontal surgery whereas the control group will receive orthodontic intervention 3 months after periodontal surgery. Supragingival scaling will be done in both the groups at 3 month intervals as per requirement.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 EARLY (Experimental): In experimental group Orthodontic treatment will be started (early) 10 days after periodontal surgery
  Interventions: Procedure: Fixed Orthodontic treatment
- Group 2 DELAYED (Experimental): control group will receive orthodontic intervention(delayed) 3 months after periodontal surgery
  Interventions: Procedure: Fixed Orthodontic treatment

INTERVENTIONS:
Procedure: Fixed Orthodontic treatment — All the patients will receive the indicated periodontal surgical treatment. and the patients will then be randomly divided into two groups - test group and control group Orthodontic treatment will be started in the test group (EARLY)10 days after periodontal surgery whereas the control group will receive orthodontic intervention (DELAYED) 3 months after periodontal surgery.

SUMMARY:
RESEARCH QUESTION: Will there be a difference in periodontal health of two groups of periodontally compromised orthodontic patients with early and delayed start of orthodontic treatment after periodontal surgery? Population: Adult orthodontic patients with periodontally compromised dentition requiring periodontal surgical management Intervention: Fixed orthodontic treatment started 10 days after periodontal surgery Control group: Fixed orthodontic treatment started 3 months after periodontal surgery Outcomes: changes in osseous (Alveolar bone level) and non-osseous (PI, GI, BOP, PD, CAL) periodontal parameters of the teeth involved in periodontal surgery.

Time frame: One year and four months Study Design: Prospective, randomized controlled clinical trial. Specific: Yes Measurable: Yes Achievable: Yes Relevant: Yes Time: One year and four months Feasible: Trained staff, infrastructure, time, study design Interesting: A new treatment protocol will be investigated. Novel: No study comparing these waiting time intervals after periodontal surgery before starting orthodontic treatment.

Ethical: Yes Relevant: As there is no clarity on waiting period after periodontally surgery in periodontally compromised adult patients, this study will be of great help in establishing treatment management protocol of such patients.

DETAILED DESCRIPTION:
Sample size: The CAL difference of 1.07 mm was considered to be of clinical importance between the test and control groups. To be able to detect a clinically meaningful difference in mean CAL of 1.0 mm between groups, standard deviation of 1.0 mm, with a power of 80% and an alpha-level at 0.05, 15 patients are needed in each group. Accounting for a 20% drop out rate 18 patients will be enrolled in each group.

Method of study: All the patients included in the study will receive a detailed periodontal evaluation and all periodontal parameters (osseous and non-osseous) will be recorded at the baseline and Phase I periodontal therapy will be provided. This will include oral hygiene instruction, scaling and root planning and re-evaluation after one weeks. If the patients are able to maintain oral hygiene after preliminary periodontal intervention they will be included in further stages of the study. All the patients will receive the indicated periodontal surgical treatment. and the patients will then be randomly divided into two groups - test group and control group Orthodontic treatment will be started in the test group 10 days after periodontal surgery whereas the control group will receive orthodontic intervention 3 months after periodontal surgery. Supragingival scaling will be done in both the groups at 3 month intervals as per requirement.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Adult patients (20-40 years) with periodontally compromised dentition indicated for periodontal surgical intervention.
* Class I malocclusion that needs orthodontic treatment.
* Stage II and Stage III periodontitis according to the criteria of 2017 world workshop.

Exclusion Criteria:

* Systemic illness known to affect the periodontium or outcome of periodontal and orthodontic therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Pregnant or lactating women.
* Smokers
* Noncompliance to oral hygiene measures after Phase I therapy.
* Presence of trauma from occlusion (TFO).
* Stage IV periodontitis according to the criteria of 2017 world workshop

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Pocket depth | T0 - baseline records, before beginning of any treatment
  measured from the gingival margin to the bottom of the pocket at six sites and recorded to the nearest millimetre
Pocket depth | T1 - 3 months post periodontal surgery
  measured from the gingival margin to the bottom of the pocket at six sites and recorded to the nearest millimetre
Pocket depth | T2 - one year after start of orthodontic treatment
  measured from the gingival margin to the bottom of the pocket at six sites and recorded to the nearest millimetre
alveolar crest bone level | Alveolar bone level will be recorded with the help of CBCT at T0 intervals.T0 - baseline records, before beginning of any treatment,
  alveolar crest bone level using cone beam computed tomography (CBCT) between the two groups, with one group beginning orthodontic treatment 10 days and the second group 3 months after undergoing periodontal surgical treatment.
alveolar crest bone level | Alveolar bone level will be recorded with the help of CBCT at T2 time intervals,T2 - one year after start of orthodontic treatment.
  alveolar crest bone level using cone beam computed tomography (CBCT) between the two groups, with one group beginning orthodontic treatment 10 days and the second group 3 months after undergoing periodontal surgical treatment.
Clinical attachment loss (CAL) | T0 - baseline records, before beginning of any treatment
  Loss of clinical attachment measured from the Cemento enamel junction to the base of pocket
Clinical attachment loss (CAL) | T1 - 3 months post periodontal surgery
  Loss of clinical attachment measured from the Cemento enamel junction to the base of pocket
Clinical attachment loss (CAL) | T2 - one year after start of orthodontic treatment
  Loss of clinical attachment measured from the Cemento enamel junction to the base of pocket

SECONDARY OUTCOMES:
Bleeding on probing, | T0 - baseline records, before beginning of any treatment
  Bleeding on probing measured at number of sites showing bleeding on using periodontal probe
Bleeding on probing, | T1 3 months post periodontal surgery
  Bleeding on probing measured at number of sites showing bleeding on using periodontal probe
Bleeding on probing, | T2 - one year after start of orthodontic treatment.
  Bleeding on probing measured at number of sites showing bleeding on using periodontal probe
Plaque index | T0 - baseline records, before beginning of any treatment
  Plaque index measured using pre specified scoring methods defined by Silness P and Loe H 1964
Plaque index | T1 3 months post periodontal surgery
  Plaque index measured using pre specified scoring methods defined by Silness P and Loe H 1964
Plaque index | T2 - one year after start of orthodontic treatment.
  Plaque index measured using pre specified scoring methods defined by Silness P and Loe H 1964
Gingival Index | T0 - baseline records, before beginning of any treatment
  Gingival index measured using pre specified scoring methods defined by Loe H and Silness P 1963
Gingival Index | T1 3 months post periodontal surgery
  Gingival index measured using pre specified scoring methods defined by Loe H and Silness P 1963
Gingival Index | T2 - one year after start of orthodontic treatment.
  Gingival index measured using pre specified scoring methods defined by Loe H and Silness P 1963

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No